CLINICAL TRIAL: NCT07372963
Title: Prospective Clinical Study and Exploration of 18F-FAPI PET/CT Imaging in Cancers of Unknown Primary Site
Brief Title: 18F-FAPI PET in Cancers of Unknown Primary Site
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: FirstZhejiangU-FAPI-CUPs
Record Dates: First submitted 2025-12-25; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Cancer of Unknown Primary Site
MeSH Terms: conditions — Neoplasms, Unknown Primary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- FAPI-cups: FAPI PET scan in patients with CUPs
  Interventions: Diagnostic Test: 18F-FAPI PET

INTERVENTIONS:
Diagnostic Test: 18F-FAPI PET — 18F-FAPI-04 PET/CT

SUMMARY:
This study aims to evaluate the diagnostic efficacy, therapeutic assessment, prognostic analysis, and impact on clinical treatment decisions of 18F-FAPI PET/CT in patients with cancer of unknown primary.

DETAILED DESCRIPTION:
Primary endpoint: Diagnostic efficacy of 18F-FAPI PET/CT in patients with undetermined primary tumor (sensitivity, specificity, accuracy).

secondary end points:

* The diagnostic performance of 18F-FAPI PET/CT compared with CT, MR and 18F-FDG PET in the clinical application of cancer with unknown primary site was compared.

  ④Assess the heterogeneity of sensitivity and specificity of 18F-FAPI PET/CT for different system sites (neck/thorax/abdomen).
* Study on efficacy evaluation and prognostic prediction of 18F-FAPI PET/CT in patients with primary tumors of unknown origin.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinical or imaging suspicion of cancer of unknown primary origin.
2. Patients with 18F FAPI PET scans.

Exclusion Criteria:

1. Concurrent presence of other active malignant tumors or a history of other malignant tumors within the past 5 years;
2. Severe uncontrollable diseases or active infections;
3. Ineligible participants for project informed consent.
4. Pregnant and lactating women.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy | through study completion, an average of 1.5 year
  Sensitivity, specificity, positive and negative predictive value of 18F-FAPI PET/CT Imaging in cancers of unknown primary site

SECONDARY OUTCOMES:
Standard uptake value （SUV）of tumor | through study completion, 3-4 years
  This measure evaluates the association between baseline 18F-FAPI PET parameters (e.g., SUVmax, SUVmean).
Metabolic tumor volume (c) and total lesion glycolysis (TLG) of tumor | through study completion, 3-4 years
  This measure evaluates the association between baseline 18F-FAPI PET parameters (MTV in cm3, TLG in cm3*SUV）
Prognostic Value of Baseline 18F-FAPI PET for Progression-Free Survival (PFS) in High-Risk Patients | through study completion, 3-4 years
  Prognostic Value of Baseline 18F-FAPI PET for Progression-Free Survival (PFS) in High-Risk Patients

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2025-10-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT07372963/ICF_000.pdf